CLINICAL TRIAL: NCT01359345
Title: The Prevalence and Severity of Nephrogenic Systemic Fibrosis in Patients Whom Underwent Imaging With Gadollinium(MRI/MRA) in University Hospital of Tehran Heart Center in 2003-2008
Brief Title: Nephrogenic Systemic Fibrosis With Gadollinum
Acronym: NSF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Imam Khomeini Hospital (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Principal Investigator, Mohammad Reza Khatami, Associate professor, Imam Khomeini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GADOLLINUM; 6553-30-04-86
Record Dates: First submitted 2009-10-26; First posted 2011-05-24 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Nephrogenic Systemic Fibrosis; Renal Failure
Keywords: NSF; ESRD; MRA; MRI; occurrence of NSF; Use of Gadollinum
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy; Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): The patients with renal failure in whom Gadollinume has being used
  Interventions: Drug: gadollinum

INTERVENTIONS:
Drug: gadollinum — use of on injection gadollinum Iv for imaging

SUMMARY:
Recently there is increasing reports of NEPHROGENIIC SYSTEMIC FIBROSIS(NSF) in patients with severe renal failure mainly in patients under dialysis in whom gadollinum is being used.

The investigators will evaluate the prevalence and severity of NSF in patients with different degree of renal failure whom underwent imaging with Gadolinum.

DETAILED DESCRIPTION:
NSF is a progressive and potentially fatal disease reported mainly in End Stage Renal Disease (ESRD) patients in whom Gadolinume been used as contrast agent. Skin is the main organ of involvement but other vital organs like myocard,lung,liver may also be involved.Gadollinum is known as a safe contrast in renal disease patients in comparison with conventional nephrotoxic radiocontrast agents,but with increasing reports of NSF with Gadollinum the use of this agent in renal failure patients is under question.

We will retrospectively evaluate the occurrence of this complication in all patients with different degree of renal failure whom underwent MRA or MRI with Gadollinum in Tehran Heart Center since 2003 till now and we will describe the severity and distribution pattern of lesions and the relation of this complication to the severity of renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Renal Failure
* Use of Gadollinum

Exclusion Criteria:

* No consent
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
occurrence of fibrosis | after 2 month of exposure with gadollinum

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Khatami, MD, Principal Investigator — TUMS
Locations (1):
- Tehran Heart Center, Tehran, Iran